CLINICAL TRIAL: NCT03262662
Title: EVarQuit: Extended Pre-quit Varenicline to Assist in Quitting Smoking
Acronym: EVarQuit
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Pfizer (Industry)
Responsible Party: Principal Investigator, Larry Hawk, Ph.D., Professor, Department of Psychology, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY00000911; R01CA206193 (NIH)
Record Dates: First submitted 2017-08-22; First posted 2017-08-25 (Actual); Results first posted 2023-07-11 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Tobacco Smoking
MeSH Terms: conditions — Tobacco Smoking | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Extended Run-In (Experimental): ** 4 weeks of varenicline prior to the target quit date (TQD) **
  + 11 weeks of post-TQD varenicline
  Standard varenicline dosing titration in initial week of therapy (one 0.5 mg tablet orally daily x 3 days, then one 0.5 mg tablet twice daily x 4 days); then 1 mg twice daily thereafter.
  Brief individual counseling at clinic visits
  Interventions: Drug: Varenicline; Behavioral: Brief smoking cessation counseling
- Standard Run-In (Active Comparator): ** 3 weeks of placebo followed by 1 week of varenicline prior to the target quit date (TQD) **
  + 11 weeks of post-TQD varenicline
  Standard varenicline dosing titration in initial week of therapy (one 0.5 mg tablet orally daily x 3 days, then one 0.5 mg tablet twice daily x 4 days); then 1 mg twice daily thereafter.
  Brief individual counseling at clinic visits
  Interventions: Drug: Varenicline; Behavioral: Brief smoking cessation counseling

INTERVENTIONS:
Drug: Varenicline — oral varenicline tablets
  Other Names: Chantix
Behavioral: Brief smoking cessation counseling — ~10-minute individual counseling at each of 6 clinic visits

SUMMARY:
Varenicline is the most effective smoking cessation therapy available. Nevertheless, most smokers using varenicline relapse within the first few months after quitting. Varenicline is hypothesized to help smokers to quit in part by reducing the reinforcing effects of smoking during the standard 1-week pre-quitting treatment phase. Learning theory and previous human and animal research support the hypothesis that a longer period of varenicline treatment prior to the target quit date (TQD) will lead to greater reductions in smoking before quitting, and higher long-term cessation rates, compared to standard varenicline treatment. Building on promising preliminary clinical data, the study tests these hypotheses with a full-scale randomized clinical trial (RCT). 320 treatment-seeking smokers will be randomized to a standard run-in group (3 weeks of placebo, followed by the standard 1 week of pre-TQD varenicline) or an extended run-in group (4 weeks of pre-TQD varenicline). Both groups will receive brief individual cessation counseling and 11 weeks of post-TQD varenicline. The primary outcome measure will be bio-verified continuous abstinence at end-of-treatment (weeks 8-11 post-quit; cessation at 26-weeks post TQD will also be examined. Hypothesized mediating mechanisms (e.g., smoking reinforcement) will be evaluated by behavioral, physiological, and subjective measures assessed both in the lab and using real-world, real-time electronic momentary assessments (EMA). The investigators predict that long-term, bio-verified smoking cessation will be improved among the extended run-in group compared to the standard run-in group. The investigators further predict the improved clinical outcomes with extended run-in varenicline will be explained (or mediated) by greater pre-quit reductions in smoking reinforcement among the extended run-in group compared to the standard run-in group. The significance of this work is clear: The project aims to make best available treatment for smoking cessation even better, using a method that is ripe for dissemination and an approach that will elucidate critical mechanisms to target in the next generation of treatment enhancement.

ELIGIBILITY:
Inclusion Criteria:

* Smoking at least 10 cigarettes per day (CPD) for the past 6 months and expired-air carbon monoxide (CO) >7 at intake. NOTE: To reduce exclusion of Black participants, the CPD criterion was reduced to 5 and the carbon monoxide criterion was eliminated in November, 2019.
* At least moderately motivated to quit smoking and intention to make a quit attempt with varenicline 1 month after treatment begins.
* Planning to remain in western New York (NY) during the study period
* Willing to use varenicline and to refrain from other cessation treatments and tobacco products during the study period.
* English speaker
* To be intent-to-treat (ITT), the participant must complete Lab Visit 1 and meet minimal completion rate for real-world (EMA) assessments.

Exclusion Criteria:

* Use of other tobacco products, including e-cigarettes, in past 7 days
* Use of smoking cessation medication, including nicotine replacement therapy, in the past 14 days
* Prior allergy/hypersensitivity to varenicline
* Pregnant or breast-feeding
* Substance use:

  * Alcohol: AUDIT score > 15 at intake, suggestive of alcohol dependence and warranting treatment; for those with scores between 8 and 15, the investigators will advise reducing drinking).
  * Medical treatment for substance use (SU) in past 3 months, including Suboxone (buprenorphine) and methadone (at phone screen)
  * Using a combination of the National Institute on Drug Abuse (NIDA) modified ASSIST (4-26 = moderate risk; 27+ = high risk) and urine toxicology screen (both at intake):

    * Cannabis: ASSIST=27+ (tox screen not used)
    * Cocaine: ASSIST=7+ OR positive tox screen
    * Methamphetamine: ASSIST=7+ OR positive tox screen
    * Inhalants, hallucinogens, sedatives, or sleeping pills: ASSIST score = 7+
    * Prescription stimulants: With prescription, ASSIST 27+; Without prescription, ASSIST 7+
    * Opioids: With prescription, ASSIST 27+ (note ineligible if prescription is for buprenorphine or methadone); Without prescription, ASSIST 7+ OR positive tox screen

(Note: ASSIST 4+ modified to 7+ in 2018 to avoid excluding people with past SU problems. clinicaltrials.gov edited 12/18/18)

* Psychiatric:

  * Antipsychotic medications
  * Lifetime history of schizophrenia or bipolar disorder
  * Evidence of current major depression (per Patient Health Questionnaire (PHQ-9) at intake
  * Past 10 years suicidal ideation (SI) / behavior. At intake, all of the following are exclusionary on the baseline Columbia-Suicide Severity Rating Scale (Posner et al., 2008): SI without intent (C-SSRS #1, #2, or #3), if any intensity rating (Frequency, Duration, Controllability, Deterrents, or Reasons for Ideation) is > 2; SI with intent (C-SSRS #4, or #5), regardless of intensity ratings; Suicidal Behavior (any suicide attempt, interrupted attempt, aborted attempt, or suicide preparatory acts or behavior on the C-SSRS).
* Any medical condition, illness, disorder or concomitant medication that compromises participant safety or treatment, as determined by the Principal Investigator and/or Study Physician.
* Inability to provide informed consent or complete any of the study tasks as determined by the Principal Investigator and/or Study Physician.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Approximately equal numbers of men and women will participate.
Enrollment: 320 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2021-04-05 (Actual); Study Completion 2021-07-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- State University of New York at Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
We plan to share study data through the NIDA-supported NAHDAP repository. IPD to be shared include baseline participant characteristics, intervention group, smoking abstinence, and adverse events.
Supporting Information: Study Protocol, ICF
Time Frame: 2023. We are currently awaiting confirmation from NAHDAP that our archival plan fits their expectations. Data will be available indefinitely (as long as NAHDAP is supported).
Access Criteria: Public release; anyone who registers on the website.

REFERENCES:
- [Derived] Cooper RK, Gass J, Mahoney MC, Tiffany ST, Colder CR, Maguin E, Schlienz NJ, Lawson SC, Tyndale RF, Sandhur B, Hawk LW. Do lab-based assessments of pretreatment smoking reinforcement and cue-specific craving predict smoking cessation with varenicline? Psychol Addict Behav. 2025 Dec;39(8):713-722. doi: 10.1037/adb0001081. Epub 2025 Jul 28. PMID 40720285
- [Derived] Tonkin S, Gass J, Wray J, Maguin E, Mahoney M, Colder C, Tiffany S, Hawk LW Jr. Evaluating Declines in Compliance With Ecological Momentary Assessment in Longitudinal Health Behavior Research: Analyses From a Clinical Trial. J Med Internet Res. 2023 Jun 22;25:e43826. doi: 10.2196/43826. PMID 37347538
- [Derived] Hawk LW Jr, Tiffany ST, Colder CR, Ashare RL, Wray JM, Tyndale RF, Brandon TH, Mahoney MC. Effect of Extending the Duration of Prequit Treatment With Varenicline on Smoking Abstinence: A Randomized Clinical Trial. JAMA Netw Open. 2022 Nov 1;5(11):e2241731. doi: 10.1001/jamanetworkopen.2022.41731. PMID 36367720
- [Derived] Ferkin AC, Tonkin SS, Maguin E, Mahoney MC, Colder CR, Tiffany ST, Hawk LW. A Psychometric Evaluation of the Stanford Expectations of Treatment Scale (SETS) in the Context of a Smoking Cessation Trial. Nicotine Tob Res. 2022 Nov 12;24(12):1914-1920. doi: 10.1093/ntr/ntac187. PMID 35906990
- [Derived] Mahoney MC, Park E, Schlienz NJ, Duerr C, Hawk LW. Transitioning to Remote Clinic Visits in a Smoking Cessation Trial During the COVID-19 Pandemic: Mixed Methods Evaluation. JMIR Form Res. 2021 Apr 30;5(4):e25541. doi: 10.2196/25541. PMID 33878020
- [Derived] Lawson SC, Gass JC, Cooper RK Jr, Tonkin SS, Colder CR, Mahoney MC, Tiffany ST, Hawk LW Jr. The impact of three weeks of pre-quit varenicline on reinforcing value and craving for cigarettes in a laboratory choice procedure. Psychopharmacology (Berl). 2021 Feb;238(2):599-609. doi: 10.1007/s00213-020-05713-7. Epub 2020 Nov 21. PMID 33219852

RESULTS

PARTICIPANT FLOW:
Groups:
- Extended Run-In: ** 4 weeks of varenicline prior to the target quit date (TQD) **
  + 11 weeks of post-TQD varenicline
  Standard varenicline dosing titration in initial week of therapy (one 0.5 mg tablet orally daily x 3 days, then one 0.5 mg tablet twice daily x 4 days); then 1 mg twice daily thereafter.
  Brief individual counseling at clinic visits
  Varenicline: oral varenicline tablets
  Brief smoking cessation counseling: ~10-minute individual counseling at each of 6 clinic visits
- Standard Run-In: ** 3 weeks of placebo followed by 1 week of varenicline prior to the target quit date (TQD) **
  + 11 weeks of post-TQD varenicline
  Standard varenicline dosing titration in initial week of therapy (one 0.5 mg tablet orally daily x 3 days, then one 0.5 mg tablet twice daily x 4 days); then 1 mg twice daily thereafter.
  Brief individual counseling at clinic visits
  Varenicline: oral varenicline tablets
  Brief smoking cessation counseling: ~10-minute individual counseling at each of 6 clinic visits
Period: Overall Study
Arm/Group | Extended Run-In | Standard Run-In
Started | 163 | 157
Retained at Wk 15 (EOT) | 127 | 126
Retained at Wk 28 (6-month Follow-up) | 124 | 121
Completed | 163 (Intent-to-treat) | 157 (Intent-to-treat)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Extended Run-In | Standard Run-In | Total
Number analyzed (Participants) | 163 | 157 | 320
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.8 (10.3) | 53.5 (10) | 53.7 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 89 | 179
  Male | 73 | 68 | 141
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8
  Not Hispanic or Latino | 159 | 153 | 312
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Self-reported race
  Participants
    Race: White/Caucasian | 122 | 118 | 240
    Race: Black/African American | 33 | 34 | 67
    Race: American Indian / Alaska Native | 1 | 2 | 3
    Race: Other | 4 | 3 | 7
    Race: More than 1 race | 2 | 0 | 2
    Race: Refused / prefer not to answer | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 163 | 157 | 320
Cigarettes per day [Mean (Standard Deviation); unit: Cigarettes per day] — Self-reported cigarettes smoked per day, on average, over the past 6 months
  Cigarettes per day | 17.9 (7.2) | 18.4 (7.3) | 18.1 (7.2)
Salivary cotinine [Mean (Standard Deviation); unit: ng/mL] — Population: Baseline cotinine data were missing for one participant in the standard run-in group.
  ng/mL
    number analyzed (Participants) | 163 | 156 | 319
    (all) | 312 (158) | 312 (164) | 312 (161)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Continuous Abstinence at End-of-Treatment (EOT) as Assessed by Self-Report and Bio-verification
Description: Number of participants with bio-verified (cotinine level of 15 ng/mL or less) self-reported continuous abstinence from smoking (not even a puff) during the final four weeks of treatment
Time Frame: Self-report Treatment Weeks 12-15; bio-verification ~Week 16
Population: Intent-to-treat analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Extended Run-In | Standard Run-In
Number analyzed (Participants) | 163 | 157
Participants | 64 | 57

2. Secondary Outcome: Pre-quit Change in Cigarettes Smoked Per Day
Description: Percent change in smoking behavior (self-reported cigarettes per day; CPD) from timeline follow-back (TLFB) interviews during the pre-quit phase of the study.
Time Frame: Treatment Week 1 vs. Treatment Week 4 (final week before TQD)
Population: This analysis is not based on ITT, as only participants with complete TLFB data for Weeks 1 and 4 were included in the analysis; early in the trial, pre-quit TLFB was not consistently obtained due to staff error.
Measure: Mean (Standard Error); unit: percent change in CPD
Arm/Group | Extended Run-In | Standard Run-In
Number analyzed (Participants) | 128 | 123
percent change in CPD | -38.8 (2.7) | -17.5 (2.8)

3. Secondary Outcome: Number of Participants With Continuous Abstinence at 6-Month Follow-Up as Assessed by Self-Report and Bio-verification
Description: Number of participants with continuous abstinence at the 6-month follow-up (no self-reported smoking during weeks 12-28 AND cotinine level 15 ng/mL or less at EOT and 6 month follow-up)
Time Frame: Self-report Treatment Weeks 12-28; bio-verification ~Week 16 and ~Week 29
Measure: Count of Participants; unit: Participants
Arm/Group | Extended Run-In | Standard Run-In
Number analyzed (Participants) | 163 | 157
Participants | 37 | 29

ADVERSE EVENTS:
Time Frame: Adverse events were assessed at intake and clinic visits which occurred across the first two months of treatment.
Description: At each visit, participants completed a 32-item symptom checklist, as in prior work.
  Suicidality was assessed at each visit with the Columbia Suicide Severity Rating Scale.
  Here, data on adverse events are reported for each of three treatment phasesphases (pre-treatment phase [intake visit & clinic visit 1); pre-quit run-in manipulation phase [clinic visits 2&3; extended run-in group taking varenicline, standard run-in group taking placebo], and early quit phase [clinic visits 4&5]).
Groups:
- Pre-Treatment Phase (Intake Visit & Clinic 1): Extended Run-In Group; Pre-Treatment Phase (Intake Visit & Clinic 1): Standard Run-In Group: Pre-Treatment Phase: Intake Visit and Clinic 1 assessments occurred prior to initiating treatment
  Brief smoking cessation counseling: ~10-minute individual counseling at each clinic visit
- Pre-Quit Run-In Manip Phase (Clinic 2 & 3): Extended Run-In Group: Pre-Quit Run-In Manipulation Phase (3 weeks):
  All participants began taking study medication following Clinic 1
  The extended run-in group took varenicline:
  Varenicline dosing titration in initial week of therapy (one 0.5 mg tablet orally daily x 3 days, then one 0.5 mg tablet twice daily x 4 days); then 1 mg twice daily thereafter.
  Brief smoking cessation counseling: ~10-minute individual counseling at each clinic visit
- Pre-Quit Run-In Manip Phase (Clinic 2 & 3): Standard Run-In Group: Pre-Quit Run-In Manipulation Phase (3 weeks):
  All participants began taking study medication following Clinic 1
  The standard run-in group took placebo.
  Brief smoking cessation counseling: ~10-minute individual counseling at each clinic visit
- Early Quit Phase (Clinic 4 & 5): Extended Run-In Group: Early Quit Phase (3 weeks):
  The extended run-in group continued varenicline, two 0.5 mg varenicline twice daily during Week 4 (to match the placebo group and maintain the blind); 1 mg twice daily thereafter.
  Brief smoking cessation counseling: ~10-minute individual counseling at each clinic visit
- Early Quit Phase (Clinic 4 & 5): Standard Run-In Group: Early Quit Phase (3 weeks)
  Varenicline dosing titration in Week 4 (one 0.5 mg tablet and 3 placebo orally daily x 3 days, then one 0.5 mg tablet and 1 placebo twice daily x 4 days); then 1 mg twice daily thereafter.
  Brief smoking cessation counseling: ~10-minute individual counseling at each clinic visit
Arm/Group | Pre-Treatment Phase (Intake Visit & Clinic 1): Extended Run-In Group | Pre-Treatment Phase (Intake Visit & Clinic 1): Standard Run-In Group | Pre-Quit Run-In Manip Phase (Clinic 2 & 3): Extended Run-In Group | Pre-Quit Run-In Manip Phase (Clinic 2 & 3): Standard Run-In Group | Early Quit Phase (Clinic 4 & 5): Extended Run-In Group | Early Quit Phase (Clinic 4 & 5): Standard Run-In Group
All-Cause Mortality (participants affected / at risk) | 0/163 | 0/157 | 0/157 | 0/147 | 0/150 | 0/146
Serious Adverse Events (participants affected / at risk) | 0/163 | 0/157 | 1/157 | 0/147 | 2/150 | 2/146
Other Adverse Events (participants affected / at risk) | 125/163 | 121/157 | 131/157 | 104/147 | 116/150 | 104/146
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pre-Treatment Phase (Intake Visit & Clinic 1): Extended Run-In Group (N=163) | Pre-Treatment Phase (Intake Visit & Clinic 1): Standard Run-In Group (N=157) | Pre-Quit Run-In Manip Phase (Clinic 2 & 3): Extended Run-In Group (N=157) | Pre-Quit Run-In Manip Phase (Clinic 2 & 3): Standard Run-In Group (N=147) | Early Quit Phase (Clinic 4 & 5): Extended Run-In Group (N=150) | Early Quit Phase (Clinic 4 & 5): Standard Run-In Group (N=146)
pyelonephritis/nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
urinary tract infection (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Scabies (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Bilateral hand swelling (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
bowel obstruction/laparotomy for lysis of adhesions (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
urinary frequency and incisional pain 3 days after elective inguinal hernia repair (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pre-Treatment Phase (Intake Visit & Clinic 1): Extended Run-In Group (N=163) | Pre-Treatment Phase (Intake Visit & Clinic 1): Standard Run-In Group (N=157) | Pre-Quit Run-In Manip Phase (Clinic 2 & 3): Extended Run-In Group (N=157) | Pre-Quit Run-In Manip Phase (Clinic 2 & 3): Standard Run-In Group (N=147) | Early Quit Phase (Clinic 4 & 5): Extended Run-In Group (N=150) | Early Quit Phase (Clinic 4 & 5): Standard Run-In Group (N=146)
Nausea (Gastrointestinal disorders) | 13 | 13 | 45 | 26 | 48 | 42
Vomiting (Gastrointestinal disorders) | 1 | 2 | 11 | 5 | 10 | 9
Abdominal Pain (Gastrointestinal disorders) | 8 | 9 | 19 | 8 | 13 | 12
Indigestion (Gastrointestinal disorders) | 17 | 13 | 13 | 6 | 10 | 9
Diarrhea (Gastrointestinal disorders) | 12 | 13 | 13 | 7 | 12 | 5
Constipation (Gastrointestinal disorders) | 16 | 11 | 22 | 23 | 25 | 28
Dry mouth (Gastrointestinal disorders) | 25 | 37 | 33 | 43 | 29 | 37
Flatulence (Gastrointestinal disorders) | 3 | 15 | 11 | 15 | 12 | 10
Gas (Gastrointestinal disorders) | 19 | 23 | 28 | 20 | 25 | 23
Agitation (Psychiatric disorders) | 37 | 31 | 32 | 26 | 29 | 41
Depressed Mood (Psychiatric disorders) | 20 | 27 | 21 | 16 | 23 | 14
Irritability (Psychiatric disorders) | 58 | 50 | 55 | 47 | 49 | 56
Hostility (Psychiatric disorders) | 9 | 2 | 10 | 5 | 11 | 6
Anxiety (Psychiatric disorders) | 36 | 34 | 26 | 25 | 25 | 32
Insomnia (General disorders) | 25 | 29 | 29 | 27 | 33 | 29
Abnormal dreams (General disorders) | 6 | 9 | 41 | 15 | 35 | 24
Other Sleep Problems (General disorders) | 23 | 29 | 25 | 14 | 22 | 15
Increased Heart Rate (Cardiac disorders) | 11 | 3 | 8 | 7 | 5 | 4
Chest Pain (Cardiac disorders) | 9 | 6 | 9 | 5 | 7 | 4
Headache (Nervous system disorders) | 39 | 47 | 31 | 39 | 26 | 29
Dizziness (Nervous system disorders) | 13 | 10 | 22 | 9 | 12 | 9
Attention Disturbance (Nervous system disorders) | 4 | 10 | 10 | 6 | 4 | 10
Fatigue (General disorders) | 39 | 43 | 28 | 33 | 28 | 32
Weakness (General disorders) | 14 | 9 | 8 | 7 | 8 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-06-30): https://cdn.clinicaltrials.gov/large-docs/62/NCT03262662/Prot_SAP_000.pdf
  • Informed Consent Form (2018-03-06): https://cdn.clinicaltrials.gov/large-docs/62/NCT03262662/ICF_001.pdf